CLINICAL TRIAL: NCT06601101
Title: Effects of Topical Insulin on Corneal Epithelium Healing After Corneal Crosslinking in Patients With Keratoconus: A Randomized Clinical Trial
Brief Title: Effects of Topical Insulin on Corneal Epithelium Healing After Corneal Crosslinking in Patients With Keratoconus
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Vitor Borges Guimaraes, MD, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 77229224.8.0000.5404; Topical Insulin (Other: Unicamp)
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Keratoconus; Cornea Disease; Eye Diseases; Wound Heal
Keywords: Topical Insulin; Crosslinking
MeSH Terms: conditions — Keratoconus; Corneal Diseases; Eye Diseases | interventions — Insulin; Methylcellulose

STUDY DESIGN:
Intervention Model Description: The participants will be distributed in blocks of four and stratified by gender: four small envelopes, two from each intervention group, will be sealed and placed in a larger envelope, totaling 10 larger envelopes. This ensures that in each block of four participants, two participants from each studied group will be included.
Who Masked: Participant, Care Provider, Investigator
Masking Description: After the assignment of interventions, the patient will be masked, and the research team conducting the postoperative examinations will also be masked. The assisting team performing the crosslinking will document in the research log which group the study participant belongs to. The researchers conducting the evaluations of the participants will only have access to this information at the end of the study for data analysis. In the case of suspected complications, an ophthalmologist independent of the cornea service will evaluate the patient and determine the most appropriate course of action.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): Insulin eye drops 50 IU/ml (1 drop every 6 hours)
  Interventions: Drug: Insulin
- Group B (Placebo Comparator): Placebo eye drops of 0.5% Methylcellulose (1 drop every 6 hours)
  Interventions: Drug: Placebo eye drops of 0.5% Methylcellulose

INTERVENTIONS:
Drug: Insulin — Insulin eye drops in the postoperative prescription for corneal crosslinking
  Arms: Group A
Drug: Placebo eye drops of 0.5% Methylcellulose — Placebo eye drops of 0.5% Methylcellulose in the postoperative prescription for corneal crosslinking
  Other Names: Placebo
  Arms: Group B

SUMMARY:
The cornea plays a fundamental role in vision, being a complex tissue essential for ocular health. In ophthalmological practice, there are situations such as corneal crosslinking, where damage to the corneal epithelium occurs. Crosslinking is a surgical procedure aimed at strengthening collagen bonds in the corneal stroma to prevent the progression of keratoconus, through the application of topical riboflavin followed by ultraviolet (UV-A) radiation. To enhance the effectiveness of riboflavin and UV-A radiation, the corneal epithelium needs to be removed, which can cause postoperative pain and discomfort, as well as increase the risk of complications such as infections, scarring, corneal opacities, perforations, and recurrent epithelial erosions. Several growth factors play a role in epithelial healing, and the discovery of insulin in the tear film and the presence of insulin and Insulin-Like Growth Factor (IGF-1) receptors in the cornea has raised the hypothesis that insulin may modulate the cornea's wound healing response. Since then, topical insulin has been used for various ocular pathologies, including dry eye disease, persistent epithelial defects, and neurotrophic ulcers. Based on this knowledge, studies have been developed, and promising results regarding the use of insulin in corneal healing have been reported, providing a scientific foundation for the realization of this project. The objective of this study is to evaluate the effect of insulin eye drops at a concentration of 50 IU/ml on epithelial healing in non-diabetic patients undergoing epithelial debridement for corneal crosslinking. To this end, a randomized, double-masked clinical trial will be conducted with two groups, one being the control group, in which researchers will compare the epithelial healing rate in mm²/h between the insulin group and the placebo group, as the primary outcome. Patients diagnosed with keratoconus and with an indication for the crosslinking procedure, will be invited to participate. As a result of the study, it is expected to assess and quantify the impact of topical insulin on epithelial defect closure in patients undergoing crosslinking, compared to placebo. Topical insulin may contribute to early epithelial defect closure, control of inflammation, and prevention of complications that could significantly impact visual quality.

DETAILED DESCRIPTION:
Patients from the Keratoconus Clinic at the Hospital das Clínicas of UNICAMP diagnosed with keratoconus who are indicated for crosslinking will be evaluated regarding visual acuity, refraction, biomicroscopy, automated keratometry (Auto Kerato Refractometer KR 8000® Alcon), Goldmann applanation tonometry, corneal specular microscopy (EM-3000® Tomey) for endothelial cell count, corneal tomography (Pentacam® HR 70900 Oculus), and corneal optical coherence tomography (SPECTRALIS® Heidelberg Engineering).

Once indicated for crosslinking, participants will be informed by the assistants of the Keratoconus Clinic about the study. Those who, after being informed about all aspects of the crosslinking procedure and the study, and sign the Informed Consent Form, will be randomly divided into two groups of equal size and stratified by gender. Group A will receive a prescription for insulin eye drops at a concentration of 50 IU/ml in a 0.5% methylcellulose vehicle, 1 drop four times a day, until complete corneal epithelial healing. Group B will receive a prescription for 0.5% methylcellulose eye drops (placebo), 1 drop four times a day, until complete corneal epithelial healing.

The corneal crosslinking will be performed according to the standardized protocol of the UNICAMP Ophthalmology Department by third-year residents, supervised by attending physicians and faculty members. The procedure will be carried out in an outpatient setting. The anesthetic technique is topical, achieved through the application of 0.4% benoxinate hydrochloride eye drops (Oxinest). A blepharostat is then placed, and 30% alcohol is applied to the corneal epithelium for 20 seconds, demarcated by an 8.0mm optical zone marker to prevent alcohol leakage. The alcohol is removed using an absorbent sponge (Merocel®), followed by thorough cleaning of the ocular surface with 0.9% sodium chloride solution. Next, the corneal epithelium in the 8.0mm region is removed using a corneal scraper, and the soaking procedure begins, consisting of the instillation of 1 drop of 0.1% riboflavin for 30 minutes at 3-minute intervals. After soaking, the cornea is exposed to UV-A radiation at 9 mW/cm² for 10 minutes, with riboflavin instilled every 2 minutes during this period. Once the procedure is completed, 1 drop of moxifloxacin hydrochloride 5.45mg/ml (Oftalmox®; Gbio) antibiotic eye drops is applied, and a silicone-hydrogel soft contact lens, Air Optix Plus Hydraglyde (Alcon), is placed.

Insulin eye drops 50 IU/ml (Eye Pharma) in Group A and placebo eye drops of 0.5% methylcellulose (Eye Pharma) in Group B will be prescribed every 6 hours to the eye that underwent the crosslinking procedure until complete corneal epithelialization occurs. Both the insulin and methylcellulose eye drops will come in identical bottles, making it impossible for the participants and the research team conducting the subsequent evaluations to distinguish between them. In addition to these medications, both groups will undergo postoperative treatment with prednisolone acetate 10mg/ml (Ster®; Genom) 1 drop every 6 hours, moxifloxacin hydrochloride 5.45mg/ml (Oftalmox®; Gbio) 1 drop every 6 hours, sodium hyaluronate 0.15% (Hyabak®; Genom) 1 drop every 4 hours, and silicone-hydrogel contact lenses (Air Optix Plus Hydraglyde; Alcon). These treatments are part of the standard postoperative care prescribed by the UNICAMP Department of Ophthalmology.

The primary outcome is the time to complete corneal epithelial healing. After epithelial healing, the silicone-hydrogel contact lens will be removed, and the antibiotic eye drop (Oftalmox®; Gbio) will be discontinued in both groups, as well as the insulin eye drop in Group A and the methylcellulose eye drop in Group B. At this point, both groups will be prescribed sodium hyaluronate 0.15% and prednisolone acetate 10mg/ml. Sodium hyaluronate, an ocular lubricant, will be continued until the 30th postoperative day, and prednisolone acetate will be tapered every 7 days following this schedule: every 8 hours; every 12 hours; every 24 hours; and discontinuation.

Third-year residents performing the procedures will not be masked, but they will not conduct postoperative follow-up and evaluation, which will be the responsibility of the research team. Participants will be masked, and the research team conducting the follow-up will also be masked. In case of any suspected complications related to the crosslinking procedure, an independent ophthalmologist from the cornea service will evaluate the patient without knowing to which group the patient belongs and will recommend the most appropriate treatment.

Postoperative visits will take place on the 1st, 2nd, and 3rd days after the crosslinking procedure. A fourth evaluation will occur on the 6th day post-procedure, with follow-ups every 48 hours until the corneal epithelium is fully healed. Typically, this period is not expected to exceed one week in either group. Subsequent follow-ups will occur on the 30th and 60th days post-procedure. This follow-up schedule is routinely performed by the UNICAMP Department of Ophthalmology.

At the 1st, 2nd, 3rd, and 6th postoperative days, the researcher responsible will document corneal status through photographs obtained using the Keratograph - OCULUS® device. If complete corneal healing has not occurred by the 6th day and further visits are needed, this documentation will also be performed. During these visits, objective factors such as ocular hyperemia and the extent of the epithelial defect will be assessed. For quantitative assessment of the epithelial defect, the photographs obtained using the Keratograph - OCULUS® will be analyzed using the ImageJ software (https://imagej.nih.gov/ij/). These visits will be carried out during the patient's routine care, lasting around 30 minutes. On the 30th postoperative day, biomicroscopy and applanation tonometry will be performed, with a duration of approximately 15 minutes. On the 60th postoperative day, visual acuity, refraction, biomicroscopy, corneal tomography, corneal optical coherence tomography, and endothelial cell count will be performed, with the visit lasting around 45 minutes. After this last visit, the patient will be referred back to the Keratoconus Clinic for standard follow-up, with decisions to be made by the UNICAMP Department of Ophthalmology.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of keratoconus, indicated for corneal crosslinking

Exclusion Criteria:

* Diabetes Mellitus
* Severe dry eye
* Limbal Stem Cell Deficiency
* Glaucoma
* Insulin or methylcellulose allergy

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Corneal Epithelial Healing Rate | 7 days
  Epithelial healing rate, measured daily using images obtained with the Keratograph - OCULUS® and analyzed using ImageJ software (https://imagej.nih.gov/ij/)

SECONDARY OUTCOMES:
Endothelial cell count | 60 days
  Endothelial cell count loss in each group, if any
Incidence of corneal haze | 60 days
  Incidence of corneal haze in each group

CONTACTS AND LOCATIONS:
Overall Officials: Monica Alves, PhD, Study Chair — State University of Campinas (Unicamp)
Locations (1):
- State University of Campinas, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No